CLINICAL TRIAL: NCT06121102
Title: Standard Pulsed Radiofrequency Versus Supervoltage Pulsed Radiofrequency Glossopharyngeal Nerve Therapy in Management of Oropharyngeal Cancer Pain: Randomized Clinical Trial.
Brief Title: Standard Pulsed Radiofrequency Versus Supervoltage Pulsed Radiofrequency Glossopharyngeal Nerve in Oropharyngeal Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Hany Magdy Danial, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2203-301-013
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Pulsed Radiofrequency; Super Voltage Pulsed Radiofrequency; Glossopharyngeal Nerve; Oropharyngeal Cancer; Pain
MeSH Terms: conditions — Oropharyngeal Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (supervoltage pulsed radiofrequency glossopharyngeal nerve block) (Experimental): Patients will receive supervoltage pulsed radiofrequency glossopharyngeal nerve block.
  Interventions: Procedure: Supervoltage pulsed radiofrequency glossopharyngeal nerve block
- Group B (standard voltage pulsed radiofrequency glossopharyngeal nerve block) (Active Comparator): Patients will receive standard voltage pulsed radiofrequency glossopharyngeal nerve block.
  Interventions: Procedure: Standard voltage pulsed radiofrequency glossopharyngeal nerve block

INTERVENTIONS:
Procedure: Supervoltage pulsed radiofrequency glossopharyngeal nerve block — Stimulation will be done using baylis generator both sensory at 50 HZ and 0.5-1.0 V (patient felt tingling at base of tongue, throat, ear and side of upper neck) and motor at 2 HZ and 1-2 V (contraction of stylopharyngeus muscle will be felt). After injecting 1 ml lidocaine 2% plus 1 ml (4 mg) Betamethasone (Diprofos) to augment analgesia and to lower impedance (usually it was 200-300 ohm due to bony proximity).Super voltage pulsed RF(60-75 volt according to patient tolerability will be done for 8 minutes with pulse width = 5 millisecond and pulse frequency of 2 HZ.
  Arms: Group A (supervoltage pulsed radiofrequency glossopharyngeal nerve block)
Procedure: Standard voltage pulsed radiofrequency glossopharyngeal nerve block — Stimulation will be done using baylis generator both sensory at 50 HZ and 0.5-1.0 V (patient felt tingling at base of tongue, throat, ear and side of upper neck) and motor at 2 HZ and 1-2 V (contraction of stylopharyngeus muscle will be felt). After injecting 1 ml lidocaine 2% plus 1 ml (4 mg) Betamethasone (Diprofos) to augment analgesia and to lower impedance (usually it was 200-300 ohm due to bony proximity).Super voltage8 pulsed RF will be done for 8 minutes with pulse width = 5 millisecond and pulse frequency of 2 HZ.
  Arms: Group B (standard voltage pulsed radiofrequency glossopharyngeal nerve block)

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of supervoltage pulsed radiofrequency glossopharyngeal nerve therapy versus standard pulsed radiofrequency in reduction of oropharyngeal cancer pain, through Visual analog scale score reduction.

DETAILED DESCRIPTION:
The glossopharyngeal nerve is the 9th cranial nerve. It has motor, sensory and parasympathetic function like trigeminal and facial nerves. It has its origin in the medulla oblongata and exits the skull via the jugular foramen, close to vagus and accessory nerves, together with the internal carotid artery and sympathetic nerves and terminates in the pharynx between the superior and middle pharyngeal constrictors, splitting into its terminal branches - lingual, pharyngeal, and tonsillar. Glossopharyngeal neuralgia is an extremely uncommon occurrence and accounts for only 0.2%-1.3% of the cases with facial pain. It usually affects the male individuals above 50-year age, and the reported incidence of glossopharyngeal neuralgia is roughly 0.8 per 100,000 persons per year. As per ICHD-3 (International Classification of Headache Disease- 3) classification, glossopharyngeal neuralgia is a disease characterized by an episodic unilateral pain, with sharp and stabbing in character, with sudden onset and cessation, in the glossopharyngeal nerve distribution (jaw angle, ear, tonsillar fossa and the base of the tongue). It also affect the pharyngeal and auricular branches of the vagus nerve. Pain is commonly aggravated by coughing, talking, and swallowing. Pain in glossopharyngeal neuralgia has a relapsing and remitting pattern. Vaso glossopharyngeal neuralgia may be associated with life-threatening cardiovascular features- syncope, hypotension, cardiac arrhythmias, in contrast to trigeminal neuralgia

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 70 Years.
* Both sexes
* American Society of Anesthesiologists (ASA) class II and III.
* Patients under pain management for oropharyngeal cancer (failed medical treatment or intolerance to the side effects of the drug).
* Visual analog scale (VAS) equal to or more than 6 cm in spite medical treatment.

Exclusion Criteria:

* Patient refusal.
* Patients with local or systemic sepsis.
* Uncorrectable coagulopathy.
* Unstable cardiovascular disease.
* History of psychiatric and cognitive disorders.
* Patients allergic to medication used.7
* Unable to lie supine.
* Local anatomical distortion (either congenital, post-surgical or post-radiotherapy) making intervention difficult and hazardous.
* Elongated styloid process > 25 mm.
* Age less than 18 year and more than 70 year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
The degree of pain | 3 months after the procedure
  Each patient will be instructed about pain assessment with the visual analog scale (VAS) score. VAS(0 represents "no pain" while 10 represents "the worst pain imaginable").
  VAS score will be measured at the following times: pre-procedure, day 1 after the procedure, 1,2,3,4 Weeks after the procedure, 2,3 Months after the procedure.

SECONDARY OUTCOMES:
Morphine consumption | 3 months after the procedure
  Morphine sulphate tablets drugs consumption will be recorded pre-procedure, day 1 after the procedure, 1,2,3,4 weeks after the procedure, 2,3 Months after the procedure.
Gabapentin consumption | 3 months after the procedure
  Gabapentin capsules drugs consumption will be recorded before the block and 1 week, 2 weeks, 3 weeks, 4weeks, 2 months and 3 months afterwards.
Patient satisfaction score | 1 month after the block
  Patient satisfaction score will be assessed as the following, how satisfied are the patient with the results of the procedure ? very satisfied = 5, somewhat satisfied = 4, neither satisfied nor dissatisfied = 3, somewhat dissatisfied = 2, very dissatisfied =1 It will be assessed at the following times: 24 hours after the block, 1,2 weeks after the block, 1month after the block
Percentage of functional improvement | 1 month after the procedure
  This is a self-reported analysis for the primary outcome after performing pain interventions. It is divided into 4 categories (0-25%)= no or minimal functional improvement, (more than 25-50%)= mild improvement, (more than 50-75%)= moderate improvement, and (more than 75-100%)= marked improvement.
Quality of life score | 12 weeks after the procedure
  Quality of life score improvement using the Flanagan quality of life scale (QOLS) ,which is a 16 -item (domain) questionnaire with each item scored from 1 to 7 points.
  The scale will be explained to the patient by the pain physician, and the total score will be calculated and recorded at the preoperative10 assessment (base line) and at postoperative weeks 2,3,4, 8 and 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.